CLINICAL TRIAL: NCT02341183
Title: Novel Therapies for Muco-Obstructive Lung Diseases: A Study of Tolerability and MCC Effect of Hypertonic Saline Delivered Via the tPAD in Patients With Chronic Bronchitis
Brief Title: Novel Therapies for Muco-Obstructive Lung Diseases: Testing the Transnasal Pulmonary Delivery Device in COPD/CB Subjects
Acronym: tPAD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Pro00057004
Record Dates: First submitted 2014-12-02; First posted 2015-01-19 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2016-05

CONDITIONS: COPD; Chronic Bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (2):
- A: Treatment order: tPAD treatment, then no treatment (Active Comparator): Subjects will receive one overnight treatment with 7% hypertonic saline administered via the tPAD device. They will then have one overnight stay without treatment.
  Interventions: Device: tPAD; Device: 7% hypertonic saline (510K approved as a device)
- B: Treatment order: no treatment, then tPAD treatment (Active Comparator): Subjects will have overnight stay w/o treatment, and one overnight treatment with 7% hypertonic saline administered via the tPAD device.
  Interventions: Device: tPAD; Device: 7% hypertonic saline (510K approved as a device)

INTERVENTIONS:
Device: tPAD — 7% NaCl administered continuously for 8 hours, overnight, via the tPAD device
Device: 7% hypertonic saline (510K approved as a device) — Subjects will receive overnight treatments of 7% HS via the tPAD device in both comparators, but in a randomly assigned order as described.

SUMMARY:
The primary objective of this study is to assess tolerability and effect of HS (hypertonic saline) delivered with the tPAD (transnasal Pulmonary Aerosol Delivery) device on mucociliary clearance (MCC) in chronic obstructive pulmonary disease/chronic bronchitis (COPD/CB) subjects. The investigators hypothesize that HS delivery via tPAD will be safe and and while, and will improve MCC.

DETAILED DESCRIPTION:
The beneficial effects of inhaled HS in CF patients (cystic fibrosis) have been well established. Concerns over safety and intolerability in patients with COPD/CB, based in part upon experiences with ultrasonic delivery devices, have limited interest in further exploring this therapeutic option. Although our clinical data suggests that HS delivered via jet nebulizer is generally well tolerated in patients with COPD/CB, our pre-clinical data suggests that cell shrinkage, the release of proinflammatory cytokines (i.e. IL-8), and transient cilia stasis is dependent upon the rate of aerosol delivery.

Slow/continuous delivery may avoid most/all of these detrimental effects while promoting an even greater cumulative ASL (airway surface liquid) volume increase. To translate these data into a feasible treatment strategy, a comfortable, quiet delivery device that can be used for long time periods (i.e. overnight) was developed to slowly deliver HS via a nasal cannula device while avoiding aerosol rain-out in the device's tubing. Use of a computational model (MPPD: Multiple-Path Particle Dosimetry V2.0) predicts that this device, which generates a 2 um MMAD aerosol particle, will achieve -5-8% lung deposition. When tuned to an output of ~0.033 ml/min, 8 hours of use is predicted to deposit a minimum of 140 mg of NaCI onto airway surfaces. This compares favorably to the estimated mass delivered via jet nebulizer in the clinically successful study of HS in CF (110 mg/day, assuming 19.75% deposition fraction with the Pari LC PLUS).

The proposed study is a single site, randomized, open label, cross-over trial designed to measure the tolerability and effect on mucociliary clearance following 7% HS delivered via tPAD for eight hours overnight to COPD/CB subjects. Comparison will be to measurements made following no treatment during an overnight stay. COPD/CB subjects meeting inclusion and exclusion criteria will be enrolled in the study. All study procedures will be conducted in the Clinical Translational Research Center (CTRC) at UNC Hospitals and the EPA building on Mason Farm Rd on the UNC Hospitals campus.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet the following criteria will be eligible for study participation:

1. Subjects aged 40 to 80 years (inclusive), and with a body mass index (BMI) < 35 kg/m2
2. Female subjects must be non-pregnant and must be either not sexually active, post-menopausal, surgically sterilized, or agree to use an appropriate "double-barrier" method (such as a diaphragm and condom); or, must currently be using a prescribed transdermal, injection, implant, or oral contraceptive during study participation
3. Subjects who are in their baseline state of health, as determined by a medical history and examination
4. Subjects who have normal lung function with a FEV1 of 30% - 80% predicted and a FEV1/FVC <70%
5. Subjects who are capable of providing written informed consent in English to participate in the study
6. Produces sputum two days per week or more, on average.
7. History of smoking cigarettes ≥ 10 pack years.

Exclusion Criteria:

Subjects will be excluded from the study according to the following criteria:

1. Subjects who use oxygen continuously or require it at night.
2. Subjects with an FEV1 < 30% or > 80% or an FEV1/FVC of ≥70% at screening.
3. Subjects who chronically require > 10mg per day of prednisone (or equivalent corticosteroid dose).
4. Subjects with a concomitant presence of congestive heart failure, active coronary syndromes, or other disease that in the opinion of the investigator would increase the risk resulting from participation.
5. Subjects with a recent change in respiratory medications, including new antibiotic or systemic corticosteroid interventions within the last 4 weeks.
6. Subjects with a history of intolerance or hypersensitivity to hypertonic saline or short acting inhaled beta agonists.
7. Subjects with significant bronchoreactivity by examination or PFT testing that, in the opinion of the investigator, would increase the risk of HS use.
8. Subjects who have had radiation exposure within the 12 months prior to study participation that would cause them to exceed Federal Regulations by participating in this study.
9. Subjects with symptomatically active, chronic or acute rhinosinusitis, or other nasal abnormality that could interfere with aerosol delivery or impact subject safety.
10. Subjects with a positive pregnancy test or who are nursing.
11. Subjects who have been diagnosed with obstructive sleep apnea.
12. Subjects who, in the opinion of the Principal Investigator, should not participate in the study.

    -

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Mucociliary Clearance Rate (MCC60) | The MCC outcome measure will be performed as quickly as possible (within 60 minutes) after overnight tPAD treatment
  The primary study outcome, MCC60, will serve as the primary descriptor of the mucociliary clearance rate. This assay will be begun as quickly as possible after competing the tPAD treatment (<60 minutes in all cases). MCC60 is derived by calculating the average rate of particle clearance observed during the first 60 minutes of the MCC scan procedure (MCC60; units = % cleared/time), using clearance values determined every 10 minutes for 60 minutes following inhalation of radiolabeled particles. Results obtained immediately after tPAD treatment will be compared to baseline values. Similarly, average clearance through other time domains (30 min, 90 min, 24 hrs), and from specific regions of interest (central lung; peripheral lung) will be reported as secondary MCC outcomes.

SECONDARY OUTCOMES:
Symptom survey | The outcome measure will be assessed after visits 1 and 3, immediately following each overnight visit (tPAD vs. no treatment)
  A customized survey of nasal, sleep, and respiratory symptoms will be administered to qualitatively assess the experience with the tPAD device.
Spirometry | Spirometry will be performed before each treatment visit (tPAD vs. no treatment) on Visit 1 and 3, and again after completing the assigned treatment, approximately 12 hours later
  For treatment visits, spirometry will be obtained before treatment and after the overnight treatment following the MCC study to assess safety of the assigned interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Scott H. Donaldson, MD, Principal Investigator — Associate Professor, Department of Medicine, Division of Pulmonary/Critical Care Medicine, UNC Chapel Hill
Locations (1):
- University of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States